CLINICAL TRIAL: NCT04120831
Title: Sequential B Cell/T Cell Therapy to Re-induce Humoral Immune TOLErance in ACPA- Positive Rheumatoid Arthritis A Prospective, Randomized Controlled Open Label Single-centre Clinical Trial in Adult Subjects With Active ACPA-positive Rheumatoid Arthritis Failing Methotrexate
Brief Title: TOLERA: Tolerance Enhancement in RA
Acronym: TOLERA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IM101-817
Record Dates: First submitted 2019-10-04; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Rituximab

STUDY DESIGN:
Intervention Model Description: This randomized, phase 2, single centre exploratory proof of concept study uses a sequential Rituximab/Abatacept treatment in ACPA positive rheumatoid arthritis. The study is composed of a non-blinded two arm design with a randomization of 1:1. A total amount of 20 ACPA positive RA patients are planned for enrolment. Duration of this study is planned for 52 weeks.
  Subjects willing to participate in the study have to sign a written informed consent prior to any study specific procedure, after being informed about the possible risks and possible benefits.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab + Abatacept + MTX (Experimental): all participants receive Rituximab. Study subjects will be randomized into one of two treatment arms (Abatacept+MTX vs MTX) following a 1:1 randomization at Visit 3, at the day of the 2nd Rituximab Infusion.
  Interventions: Drug: Abatacept Injection
- Rituximab + MTX (standard of care) (Active Comparator): all participants receive Rituximab. Study subjects will be randomized into one of two treatment arms (Abatacept+MTX vs MTX) following a 1:1 randomization at Visit 3, at the day of the 2nd Rituximab Infusion.
  Interventions: Drug: Abatacept Injection

INTERVENTIONS:
Drug: Abatacept Injection — Drug
  Other Names: Rituximab

SUMMARY:
Although anti-citrullinated protein antibodies (ACPA) including anti-CCP2 antibodies are known to promote inflammation and joint destruction in patients suffering from ACPA-positive rheumatoid arthritis, there are currently no therapies available to efficiently eliminate autoantibody production and to re-induce immune tolerance in these patients. However, both a B cell-targeting therapy (Rituximab) and a T cell targeting therapy (Abatacept) were described to lower anti-CCP2 antibody levels and occasionally trigger disappearance of these autoantibodies (sero conversion). By sequentially combining Rituximab and Abatacept, we thus aim to enhance the tolerogenic potential of these drugs and seek to eliminate autoantibody production and significantly lower ACPA titers. This would for the first time correspond to a "deep" immunological remission and a re-induction of immune tolerance.

DETAILED DESCRIPTION:
Based on fact that both a B cell-targeting therapy with Rituximab and a T cell-targeting therapy with Abatacept affect ACPA levels and can occasionally induce seroconversion and an immunological remission as well immune tolerance in ACPA-positive RA patients, we conclude that T/B cell-mediated autoimmunity can be in principle reversed in RA patients suffering from active disease. We hypothesize that we can increase the tolerance-inducing potency of Rituximab and Abatacept by combining these two approaches and delivering a sequential B cell/T cell therapy with Rituximab and Abatacept. Such a combined approach might increase the rate of seroconversions in RA patients and thus re-induce tolerance in a significant number of patients which would pave the way for a long-lasting "deep immunological" and drug-free remission.

In the proposed project, we thus plan to perform a sequential treatment with initial B cell depletion with Rituximab followed by blockade of the immunological synapse by Abatacept. Such an approach aims to deplete autoreactive B cells and plasmablasts, which constitute the major source for ACPA (3) and thus reboot part of the immune system, before blocking the immunological synapse in order to enable reconstitution of self-tolerance.

Based on their recently discovered pathogenic properties and to determine a potential immunological remission in the participating RA patients, we primarily plan to evaluate the effect of a sequential Rituximab/Abatacept treatment on changes in the levels of anti CCP2 antibodies between Baseline and Week 52 and will determine the rate of seroconversions.

Secondary, we plan to perform an additional quantitative and qualitative analysis of the ACPA response. Glycosylation of ACPA was shown to modulate their inflammatory activity and is thus considered to control the onset of arthritis in ACPA-positive individuals (9). We will therefore measure glycosylation (galactosylation, fucosylation and sialylation) of ACPA and total IgG. Moreover, we plan to determine changes in total IgG, IgA and IgM subclasses, numbers of total B cells and plasmablasts as well as of CCP2-specific B cells and plasmablasts in the peripheral blood of the participating patients. The clinical outcome will be measured at week 52 described by disease activity parameters and patient questionnaires.

The longitudinal setup of this proof of concept mode of action study is to evaluate the efficacy of a subsequent Abatacept therapy post B cell depletion in regard to ACPA seroconversion, ACPA titers and B cell phenotype changes.

ELIGIBILITY:
Main inclusion criteria:

Patients eligible for inclusion in this study have to fulfil all of the following criteria:

1. Understand and voluntarily sign an informed consent form
2. Male or female, age ≥ 18 years at time of consent
3. Able to adhere to the study visits and protocol
4. Satisfy the ACR-EULAR criteria of Rheumatoid Arthritis at diagnosis
5. SDAI≥11 at Screening
6. ACPA positive (anti CCP2 antibody compulsory at screening) (+/- rheumatoid factor)(≥ 40 RE/ml for CCP2 )
7. Completed vaccination for pneumococcus pneumoniae according to local guidelines at Baseline
8. Inadequate treatment response with highest tolerated dose after 3 months therapy and/or intolerance to cDMARDs specifically Methotrexate, Sulfasalazine, Hydroxychloroquine and Leflunomide or bDMARDs specifically TNF-alpha inhibitors or IL-6 receptor blockers.
9. Sulfasalazin, Hydroxychloroquine and Leflunomide must be stopped during screening phase and be replaced by Methotrexate. Leflunomide must be washed out until Baseline (Colestyramine 3x/day 8g/day for 11 days).
10. Only simultaneous therapy with Methotrexate
11. Maximum Glucocorticoid dose at Baseline: 20mg Prednisolone equivalent daily
12. JC-Virus antibody IgG and IgM in Serum negative at screening

    Main exclusion criteria:
13. Planned or ongoing pregnancy status or breast-feeding
14. Ongoing or previously treatment with Abatacept or Rituximab
15. Hypersensitivity to the active substance, mouse proteins (Rituximab), chinese hamster ovary cells (Abatacept) or other components
16. Use of any other biologic immunomodulatory agent (monoclonal antibody) except insulin.
17. Active ongoing inflammatory diseases other than RA that might confound the evaluation of the benefit of the therapy (including SLE, PSS, MCTD, SpA, Behcet disease, vasculitis or autoimmune hepatitis)
18. History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold test. If presence of latent tuberculosis is established then treatment according to local country guidelines must have been initiated but patient cannot take part in the study.
19. Known active or past infection with hepatitis B or hepatitis C at screening or baseline as defined by Antibody positivity and/or positive DNA/RNA levels of hepatitis B/C
20. Uncontrolled severe concomitant disease (including diabetes with plasma glucose >11.1 mmol/l rsp. 200 mg/dl, heart insufficiency >= NYHA III, COPD with severity >= GOLD 3, asthma according to GINA classification >= step 3)
21. Patients with weakened immune system defined as diagnosis of CVID, HIV and or total IgG levels lower than 600 mg/dl)
22. Requirement for immunization with live vaccine during the study period or within 4 weeks preceding baseline.
23. Contraindication for Rituximab or Abatacept treatment according to their SmPCs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | week 52
  Proportion of anti CCP2 antibody seroconversions in anti-CCP2-positive

SECONDARY OUTCOMES:
secondary endpoints | week 52
  Explorative serological biomarkers:
  * Change in anti CCP2 antibody levels (RE/ml)
  * Change in anti CCP2 antibodies in HLA-defined subgroups
  * Change in levels of total IgG, IgG subclasses, IgA and IgM
  * Glycosylation profile of total IgG, and of ACPA
  * Change in B cell numbers
  * Change in CCP2-specific B-cell numbers
  Clinical outcome:
  * Number of patients in DAS28, SDAI and ACR-EULAR Boolean remission at week 52
  * DAS28 , SDAI, CDAI, CRP and ESR change over 52 weeks
  * Response: ACR20, 50, 70 response at week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Universitiy Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No